CLINICAL TRIAL: NCT01679106
Title: The Effects of Continuous Transversus Abdominis Plane (TAP) Catheters on Postoperative Pain After Renal Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed because of low enrolment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-559
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Pain
Keywords: renal transplant; flank incision
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl IV PCA and placebo TAP catheter (Placebo Comparator): Patients will receive Fentanyl IV PCA and placebo TAP catheter.
  Interventions: Other: Fentanyl IV PCA and placebo TAP catheter
- TAP catheter with continuous infusion of Ropivicaine (Active Comparator): Patients will receive TAP catheter with continuous infusion of Ropivicaine for up to 48 hours after surgery.
  Interventions: Other: TAP catheter with Ropivicaine

INTERVENTIONS:
Other: TAP catheter with Ropivicaine — Patients will receive TAP catheter with continuous infusion of Ropivicaine.
  Arms: TAP catheter with continuous infusion of Ropivicaine
Other: Fentanyl IV PCA and placebo TAP catheter — Patients will receive placebo TAP catheter with Fentanyl IV PCA.
  Arms: Fentanyl IV PCA and placebo TAP catheter

SUMMARY:
Up to 174 patients undergoing renal transplantation will be randomized to one of two groups. Randomization will be based on computer-generated codes using random block sizes ranging from 4 to 8.

Group 1: TAP catheter with continuous infusion of Ropivicaine Group 2: Fentanyl IV PCA

The TAP catheter will be removed 48 hours postoperatively. Following removal, the pain scores will be assessed at 60 and 72 hours postoperatively to determine any prolonged analgesic benefit. In addition, the presence of any pain at the incision site will be noted at the 1 month surgical follow-up to determine any evidence of chronic pain.

The investigators hypothesis is that unilateral kidney transplant patients with a continuous TAP catheter will have decreased pain scores and opioid usage compared to those receiving standard analgesic therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient is >18 years of age
* The patient has provided written informed consent and understands the explanation of the protocol.
* The patient is scheduled to have a unilateral renal transplant with a flank incision

Exclusion Criteria:

* Patients aged <18.
* Patients with a known allergy to amide local anesthetics or para-aminobenzoic acid.
* Patients who are unable to understand the verbal analog pain scale.
* Patients who decline participation.
* Patients with a midline abdominal incision.
* Combined transplants, ie. Kidney-pancreas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effect of continuous TAP analgesia and pain scores | day 1
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of TAP analgesia and opioid requirements | Day 1
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of continuous TAP analgesia on pain scores | Day 2
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
effect of continuous TAP analgesia on pain scores | Day 3
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of continuous TAP analgesia on pain scores | 30 days
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of TAP analgesia on opioid requirements | Day 2
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of TAP analgesia on opioid requirements | Day 3
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).
Effect of TAP analgesia on opioid requirements | Day 30
  The primary objective is to evaluate the influence of a continuous TAP analgesia on postoperative analgesia (as defined by pain scores and opioid requirements) in patients undergoing renal transplantation, compared to standard analgesic management (IV PCA).

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Farag, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States